CLINICAL TRIAL: NCT04841538
Title: An Open-label, Multicenter, Multicohort Phase 1b/2 Clinical Trial of ES101 in Patients With Advanced Malignant Thoracic Tumors
Brief Title: A Study of ES101 (PD-L1x4-1BB Bispecific Antibody) in Patients With Advanced Malignant Thoracic Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's clinical development strategy adjustment
Sponsor: Elpiscience Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES101-2001
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Thoracic Tumors; Non-small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: ES101; INBRX-105; PD-L1; 4-1BB; PD-L1×4-1BB; PDL1; 41BB; Thoracic Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Thoracic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): ES101 is administered via intravenous infusion, 0.3mg/kg，once every 14 days, every 28 days as a treatment cycle.
  Interventions: Drug: ES101
- Cohort 2 (Experimental): ES101 is administered via intravenous infusion, 1mg/kg，once every 14 days, every 28 days as a treatment cycle.
  Interventions: Drug: ES101
- Cohort A1 (Experimental): ES101 is administered via intravenous infusion, RP2D (to be determined)，once every 14 days, every 28 days as a treatment cycle.
  Interventions: Drug: ES101
- Cohort A2 (Experimental): ES101 is administered via intravenous infusion, RP2D (to be determined)，once every 14 days, every 28 days as a treatment cycle.
  Interventions: Drug: ES101
- Cohort B (Experimental): ES101 is administered via intravenous infusion, RP2D (to be determined)，once every 14 days, every 28 days as a treatment cycle.
  Interventions: Drug: ES101
- Cohort C (Experimental): ES101 is administered via intravenous infusion, RP2D (to be determined)，once every 14 days, every 28 days as a treatment cycle.
  Interventions: Drug: ES101

INTERVENTIONS:
Drug: ES101 — The active ingredient of ES101 is a recombinant, humanized, bispecific IgG antibody that targets the human programmed death-ligand 1 (PD-L1) receptor and the human 4-1BB receptor.

SUMMARY:
The purpose of this study is to evaluate the safety, RP2D and PK/pharmacodynamic profile of ES101 monotherapy in patients with advanced NSCLC and to further evaluate the antitumor efficacy of ES101 in advanced malignant thoracic tumors, including NSCLC and SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent form.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* At least one measurable lesion is required (RECIST v1.1)
* Phase 1b: Subjects with pathologically or cytologically confirmed recurrent or metastatic NSCLC without known EGFR mutation and ALK and ROS1 gene rearrangements.
* Phase II: Subjects with pathologically or cytologically confirmed recurrent or metastatic malignant thoracic tumours who have received 1-2 lines of systemic anti-tumour therapy, including platinum regimens, and have failed, including at least 2 cycles of chemotherapy.

Exclusion Criteria:

* Prior exposure to 4-1BB agonists.
* Receipt of any anticancer investigational product or any approved drug(s) or biological products (except hormone-replacement therapy, testosterone or oral contraceptives) within 4 weeks prior to the first dose of study drug. Previous exposure to oral fluorouracils or small molecular targeted drugs require a minimum washout period of 2 weeks or 5 half-lives prior to the first dose of study drug (whichever is longer). Previous exposure to mitomycin C or nitrosourea requires a minimum washout period of 6 weeks prior to the first dose of study drug.
* Receipt of PD-L1 therapy within 24 weeks prior to the first dose of study drug.
* Known allergies to CHO-produced antibodies, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to ES101.
* Grade ≥ 3 immune-related adverse events (irAEs) or irAE that lead to discontinuation of prior immunotherapy. Some exceptions as defined per protocol apply.
* Subject has not recovered from all AEs of previous anticancer therapies to baseline or ≤ Grade 1 per CTCAE v5.0 before teh first dose of study drug. Certain exceptions as defined in protocol apply.
* Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications. Certain exceptions as defined in protocol apply.
* Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
* Systemic anti-infectious drug treatments within 4 weeks prior to the first dose of study drug.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Frequency and severity of adverse events of ES101 | 1-2 years
  Adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Phase 1b: Recommended Phase 2 Dose (RP2D) of of ES101 | 6 months
  RP2D of ES101 will be determined.
Phase 2: Objective response rate (ORR) | 2-3 years
  Tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1).

SECONDARY OUTCOMES:
Anti-tumor activity of ES101 | 2-4 years
  Tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1).
PK profile of ES101 | 2-4 years
  Assess the relationship between ES101 exposure and efficacy/adverse events.
Immunogenicity of ES101 | 2-4 years
  Frequency of anti-drug antibodies (ADA) against ES101 will be determined.
Pharmacodynamic markers | 2-4 years
  Assess PD-L1 receptor occupancy and cytokines
PD-L1 expression | 2-4 years
  Assess PD-L1 expression status of tumor tissues

IPD SHARING:
Plan to Share IPD: No